CLINICAL TRIAL: NCT00260624
Title: Escitalopram in the Treatment of Patients With Agitated Dementia
Brief Title: Escitalopram Treatment of Patients With Agitated Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP MD 43
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Alzheimer's Disease; Psychomotor Agitation
Keywords: agitation; dementia; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Dementia | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram (Lexapro)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of escitalopram (Lexapro) using 10 or 20 mg daily in patients with Alzheimer's disease who are also experiencing agitation.

DETAILED DESCRIPTION:
This study is designed for men and women over 60 who have an established diagnosis of mild to severe Alzheimer's disease and who also present behaviors of agitation such as restlessness, physical aggression, yelling and socially inappropriate interactions. While nonpharmacologic interventions are preferable, many times they are not effective alone. Each consented subject will be enrolled in a 12 week study with escitalopram, 10 or 20 mg per day. Each subject will be evaluated using rating scales designed for symptoms of Alzheimer's and agitated behavior. Each subject will also undergo physical and neurological examinations, laboratory tests and monitoring of side effects of escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Dementia of Alzheimer's type with behavioral disturbance
* Mild to severe cognitive impairment
* Age over 60
* Medically stable
* Agitation present both at screening and baseline
* Agitation not responsive to simple nonpharmacologic interventions and lasting at least 2 weeks prior to enrollment.
* Available Health Care Proxy or other legal representative to give informed consent, and patient assent.
* No planned change in environment for duration of study
* At least one reliable caregiver

Exclusion Criteria:

* Any intercurrent medical problem that could explain the agitation
* History of major depression or bipolar preceding the onset of dementia
* Other major psychiatric illness preceding the onset of dementia or mental retardation
* Other dementias
* History of alcohol abuse or dependence in the last 2 years
* Delirium (or history of delirium in the last 8 weeks)
* Treatment with other psychotropic drugs except those permitted in the protocol. Patients already treated for agitation with psychotropic medication must be able to successfully discontinue it and tolerate a washout period of no less than 1 week.
* Treatment with non-psychotropic, centrally active drugs believed to contribute to patient's agitation.
* Severe psychiatric symptoms requiring psychiatric hospitalization or suicidal, homicidal potential.
* History of intolerance to citalopram
* Noncompliance with oral medication or inability to take oral medication
* Modified Hachinski score of 4 or greater

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Agitation factor on the Neurobehavioral Rating Scale (NBRS)

SECONDARY OUTCOMES:
Total NBRS scores
Cohen-Mansfield Agitation Inventory
Neuropsychiatric Inventory
Global Clinical Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Leibovici MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Fairport Baptist Home, Fairport, New York
  - The Highlands at Brighton, Rochester, New York
  - University of Rochester, Rochester, New York